CLINICAL TRIAL: NCT02891746
Title: The Neonatal Microbiome and Its Influence on the Post-partum Period
Brief Title: Maternal and Neonatal Microbiome
Status: Withdrawn | Type: Observational
Why Stopped: recent publications have made this study obsolete
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: Mat-Neo-Micro-HMO-CTIL
Record Dates: First submitted 2016-05-31; First posted 2016-09-07 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-07

CONDITIONS: Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Premature infants: premature infants ≤ 34 weeks of gestation
  Interventions: Other: non invasive sampling
- Term infants: neonates ≥ 37 weeks gestation
  Interventions: Other: non invasive sampling

INTERVENTIONS:
Other: non invasive sampling

SUMMARY:
The aim of the study is to characterize and monitor the microbiome of premature infants born in the investigators facility until discharge from the NICU. The investigators will also examine the relationship between mode of delivery and the microbiome of the infant, while exploring various possible factors that may affect it. In addition, the investigators will compare the microbiome of premature infants to the microbiome of term babies born at the same time in the same facility.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants ≤ 34 weeks of gestation admitted to the Neonatal Intensive Care Unit at Hadassah University Hospital, Mount Scopus and their mothers.

The control group:

* Neonates ≥ 37 weeks gestation of which 50 were delivered vaginally and 50 by Caesarean section at Hadassah University Hospital, Mount Scopus and their mothers.

Exclusion Criteria:

* Neonates with congenital anomalies or metabolic conditions.

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 100 premature infants ≤ 34 weeks of gestation admitted to the Neonatal Intensive Care Unit and their mothers.
  The control group :
  100 neonates ≥ 37 weeks gestation of which 50 were delivered vaginally and 50 by Caesarean section and their mothers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Definition the flora comprising the microbiome of premature and term babies | birth

SECONDARY OUTCOMES:
Difference in the microbiome of the infants born vaginally and via caesarian section | birth
Change in the flora that constitutes the microbiome of premature babies | birth until adjusted age of 40 weeks gestation

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hadassah Medical Organization, Jerusalem, Israel, Jerusalem
  - Hadassah Medical Organization, Jerusalem

IPD SHARING:
Plan to Share IPD: Undecided